CLINICAL TRIAL: NCT03768323
Title: A Randomized Controlled Trial of Varying Airtime Incentive Amounts to Improve Interactive Voice Response (IVR) Survey Performance in Bangladesh and Uganda
Brief Title: Airtime Incentive Amounts to Improve Interactive Voice Response Surveys in Bangladesh and Uganda
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Johns Hopkins Bloomberg School of Public Health (Other)
Collaborators: The Bloomberg Family Foundation, Inc. (Other); Makerere University (Other); Institute of Epidemiology, Disease Control and Research (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: 00007318
Record Dates: First submitted 2018-08-01; First posted 2018-12-07 (Actual); Last update posted 2018-12-10 (Actual); Status verified 2018-12

CONDITIONS: Surveys and Questionnaires; Noncommunicable Diseases
Keywords: mobile phone surveys; interactive voice response; incentive
MeSH Terms: conditions — Noncommunicable Diseases

STUDY DESIGN:
Intervention Model Description: Participants were randomized to one of three airtime incentive amounts: 1) no incentive; 2) 1X incentive; or 3) 2x incentive where X was equal to 50 Bangladeshi Taka ($0.60 USD) or 5000 Ugandan Shillings (UGX; $1.35 USD as of April 3, 2018). Airtime incentives were sent if participants completed the noncommunicable disease risk factor survey
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Control (No Intervention): No airtime incentive was given for completing the survey
- 1X incentive (Experimental): 1X airtime incentive
  Interventions: Other: 1X airtime incentive
- 2X incentive (Experimental): 2X airtime incentive
  Interventions: Other: 2X airtime incentive

INTERVENTIONS:
Other: 1X airtime incentive — an incentive given in the form of airtime to motivate participants to complete the survey. Participants were given 50 Bangladeshi Taka ($0.60 USD) or 5000 Ugandan Shillings (UGX; $1.35 USD as of April 3, 2018) worth of airtime for completing the survey
  Arms: 1X incentive
Other: 2X airtime incentive — an incentive given in the form of airtime to motivate participants to complete the survey. Participants were given 100 Bangladeshi Taka ($1.20 USD) or 10000 UGX ($2.70 USD) worth of airtime for completing the survey
  Arms: 2X incentive

SUMMARY:
This study evaluates the effect of two different airtime incentive amounts on interactive voice response (IVR) survey cooperation, response, refusal, and contact rates, as compared to control group, in Bangladesh and Uganda.

DETAILED DESCRIPTION:
Using random digit dialing sampling techniques, the investigators randomized random digit dialed (RDD) participants to one of three airtime incentive amounts contingent on them completing the noncommunicable disease risk factor survey. This mobile phone survey was sent as an interactive voice response (IVR). In IVR surveys, participants use their touch tone key pad to answer pre-recorded questions. (i.e. If you are male, press 1; If you are female, press 2). This study was conducted in both Bangladesh and Uganda

ELIGIBILITY:
Inclusion Criteria:

* Access to a mobile phone
* Greater or equal to 18 years of age
* In Bangladesh, conversant in either English or Bangla language. In Uganda, conversant in either Luo, Luganda, Runyakitara, or English Languages

Exclusion Criteria:

* Less than 18 years of age

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 4233 (Actual)
Dates: Start 2017-03-26 (Actual); Primary Completion 2017-07-14 (Actual); Study Completion 2017-07-14 (Actual)

PRIMARY OUTCOMES:
Cooperation Rate #1 | Through study completion, an average of one month
  As defined by American Association for Public Opinion Research,the number of complete interviews divided by the sum of complete interviews, partial interviews, refusals, and breakoffs
Response Rate #4 | Through study completion, an average of one month
  As defined by American Association for Public Opinion Research,the number of complete and partial interviews divided by the sum of complete interviews, partial interviews, refusals, breakoffs, and the estimated eligible proportion of unknowns

SECONDARY OUTCOMES:
Refusal Rate #2 | Through study completion, an average of one month
  As defined by American Association for Public Opinion Research,the number of refusals and break-offs divided by the number of complete interviews, partial interviews, refusals, breakoffs, and the estimated eligible proportion of unknowns
Contact Rate #2 | Through study completion, an average of one month
  As defined by American Association for Public Opinion Research,the number of complete and partial interviews, refusals and break-offs divided by the number of complete interviews, partial interviews, refusals, breakoffs, and the estimated eligible proportion of unknowns

CONTACTS AND LOCATIONS:
Overall Officials: Adnan A Hyder, Phd, MBBS, Principal Investigator — Johns Hopkins Bloomberg School of Public Health; George W Pariyo, PhD, Principal Investigator — Johns Hopkins University Bloomberg School of Public Health
Locations (2):
- Institute of Epidemiology Disease Control and Research, Dhaka, Bangladesh
- Makerere University School of Public Health, Kampala, Uganda

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Gibson DG, Pariyo GW, Wosu AC, Greenleaf AR, Ali J, Ahmed S, Labrique AB, Islam K, Masanja H, Rutebemberwa E, Hyder AA. Evaluation of Mechanisms to Improve Performance of Mobile Phone Surveys in Low- and Middle-Income Countries: Research Protocol. JMIR Res Protoc. 2017 May 5;6(5):e81. doi: 10.2196/resprot.7534. PMID 28476729
- [Background] Gibson DG, Pereira A, Farrenkopf BA, Labrique AB, Pariyo GW, Hyder AA. Mobile Phone Surveys for Collecting Population-Level Estimates in Low- and Middle-Income Countries: A Literature Review. J Med Internet Res. 2017 May 5;19(5):e139. doi: 10.2196/jmir.7428. PMID 28476725
- [Background] Gibson DG, Farrenkopf BA, Pereira A, Labrique AB, Pariyo GW. The Development of an Interactive Voice Response Survey for Noncommunicable Disease Risk Factor Estimation: Technical Assessment and Cognitive Testing. J Med Internet Res. 2017 May 5;19(5):e112. doi: 10.2196/jmir.7340. PMID 28476724
- [Background] Hyder AA, Wosu AC, Gibson DG, Labrique AB, Ali J, Pariyo GW. Noncommunicable Disease Risk Factors and Mobile Phones: A Proposed Research Agenda. J Med Internet Res. 2017 May 5;19(5):e133. doi: 10.2196/jmir.7246. PMID 28476722
- [Derived] Gibson DG, Wosu AC, Pariyo GW, Ahmed S, Ali J, Labrique AB, Khan IA, Rutebemberwa E, Flora MS, Hyder AA. Effect of airtime incentives on response and cooperation rates in non-communicable disease interactive voice response surveys: randomised controlled trials in Bangladesh and Uganda. BMJ Glob Health. 2019 Sep 6;4(5):e001604. doi: 10.1136/bmjgh-2019-001604. eCollection 2019. PMID 31565406